CLINICAL TRIAL: NCT03368690
Title: Effects of Polyphenolic Extract From Pine Bark on the Inattention and Hyperactivity in Patients With Attention Deficit Hyperactivity Disorder Based on the Antioxidative Status.
Brief Title: Therapeutic Effects of Pine Bark Extracts in Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N201706026
Record Dates: First submitted 2017-08-14; First posted 2017-12-11 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-06

CONDITIONS: ADHD
Keywords: pine barkextract, antioxidant, ADHD, catecholamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligopin® (Experimental): Dietary supplement, Polyphenolic extract from pine bark. This group receives a nutritional supplement for a period of 10 weeks.
  Children and adolescent 20-50 kg body weight: 25 mg Oligopin®/day; > 50 kg body weight: 50 mg Oligopin®/day Adults 40-60 kg body weight: 100 mg Oligopin®/day; > 60 kg body weight: 150 mg Oligopin®/day
  Interventions: Dietary Supplement: Oligopin®
- Placebo (Placebo Comparator): Placebo treatment ( identical capsules containing maltodextrin and magnesium stearate )
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oligopin® — At the treatment period (0th to 4th week of the experiment), subjects with ADHD will receive 1~3 capsules of polyphenolic extract from pine bark (25mg or 50 mg Oligopin per capsule) according to their body weight and age. The 5th to 6th week will be the washout period. The control group and Oligopin group will be cross-over at 7th week to 10th week of the experiment.
  Arms: Oligopin®
Other: Placebo — At the treatment period (0th to 4th week of the experiment), subjects with ADHD will receive 1~3 capsules of polyphenolic extract from pine bark (25mg or 50 mg Oligopin per capsule) according to their body weight and age. The 5th to 6th week will be the washout period. The control group and Oligopin group will be cross-over at 7th week to 10th week of the experiment.
  Arms: Placebo

SUMMARY:
In this study, the investigators will investigate the effects of polyphenolic extract from pine bark on the inattention and hyperactivity in patients with attention deficit hyperactivity disorder (ADHD) based on antioxidative status.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a disorder characterized by developmentally inappropriate levels of impulsive behavior, hyperactivity and/or inattention. It is one of the most prevalent chronic pediatric neurodevelopmental conditions. The pathology of ADHD may relate to the oxidative stress caused by abnormal neurotransmitters. Therefore, we would like to intervene pine bark extract (PE) which can improve the symptom of inattention and hyperactivity from the psychological assessment and antioxidative status.

20 children and adolescent aged above 7 but under 20 years old and 20 adults aged from 20 to 65 years old with ADHD will be enrolled in this randomized, double-blind, cross-over and placebo controlled 10-weeks period experiment.

At the treatment period (0th to 4th week of the experiment), children and adolescent with ADHD will receive 1~2 placebo or capsules of polyphenolic extract from pine bark (25mg Oligopin per capsule) according to their body weight. On the other hand, adult with ADHD will receive 2~3 placebo or capsules of polyphenolic extract from pine bark (50mg Oligopin per capsule). The 5th to 6th week will be the washout period. The control group and Oligopin group will be cross-over at 7th week to 10th week of the experiment. Psychiatric examination and nutrition status evaluation will be carried out in this study. At the beginning, 4th, 7th and 10th week of the study, basic psychiatric examination will be carried out by clinical psychologist. Routine laboratory parameter including liver function, kidney function, lipid profile, antioxidative status and iron status will be investigated at the beginning, 4th and 10th week of the study. The nutrition status evaluation including food frequency questionnaire and three-day dietary record (two days on weekdays, one day on holiday). The food frequency questionnaire will be performed at the beginning, 4th, 7th and 10th of the experiment while three-day dietary record will be performed at 2th, 4th , 8th and 10th of the experiment. We expect that polyphenolic extract from pine bark may improve oxidative status which in turn ameliorate the attention and emotional stability in patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Children or adolescent with attention deficit hyperactivity disorder (ADHD) whose age reach 7 but under 20 and were not treated with ADHD drugs, antihypertensive drugs and dietary supplements more than 4 weeks.
2. Adults with attention deficit hyperactivity disorder (ADHD) aged from 20 to 65 and were not treated with antihypertensive drugs and dietary supplements more than 4 weeks.

Exclusion Criteria:

1. Children or adolescent treated with ADHD drugs, antihypertensive drugs and dietary supplements
2. Adults treated with antihypertensive drugs and dietary supplements
3. Nervous system diseases (including brain or other central nervous system diseases, e.g. epilepsy)
4. Autism spectrum disorder
5. Intellectual disability
6. Other mental disorders (e.g. Schizophrenia, Bipolar Disorder, Major depressive disorder, Anxiety Disorder, Personality disorders, Conduct disorder, Tourette Syndrome.)
7. Hepatic, renal, gastrointestinal and cardiovascular disorders
8. Biochemical abnormality

Ages: 7 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) | at the start of the experiment and at the 4th, 7th and 10th week
  It is used to evaluate the inattention, impulsivity and hyperactivity for children and adolescent with ADHD as rated by parents and teachers. When Inattention/Hyperactivity-impulsivity subscales approach P85, the participants are going to the next steps.
  When subjects took Oligopin that scores decrease significantly than beseline on inattention.
Adult ADHD Self-Report Scale-V1.1 (ASRS-V1.1) or Individual Subjective Perception Job Stress Scale (ISPJSS) | at the start of the experiment and at the 4th, 7th and 10th week
  It is used to evaluate the inattention, impulsivity and hyperactivity for adult with ADHD as rated by participants. The scores of ASRS-V1.1 more than 17, that can be going to the next steps.
  When subjects took Oligopin that scores decrease significantly than beseline on impulsivity and hyperactivity.
Conners' Continuous Performance Test (CPT-III) | at the start of the experiment and at the 4th, 7th and 10th week
  It is used to evaluate the inattention, impulsivity and vigilance for subjects with ADHD. T-score > 60 approach clinical standard.
  In the part of inattention, during supplementation of PE all sub-items were no difference when compared with baseline and sub-items of commissions were lower than placebo group (p<0.05). Hyperactivity results were the same with part of inattention.
Wechsler Memory Scale , WMS-III | at the start of the experiment and at the 4th, 7th and 10th week
  Use Wechsler memory test to evaluate performance progressing in concentration and impulse control for adults
  Among the result of WMS, there were no significant difference in each period.
Wisconsin Card Sorting Test, WCST | at the start of the experiment and at the 4th, 7th and 10th week
  Use Wisconsin card test to evaluate performance progressing in concentration, impulse control for adults
  Among the results of WCST, there were no significantly difference between each group.

SECONDARY OUTCOMES:
Liver function | at the start of the experiment and at the 4th, 10th week
  Serum AST,ALT and bilirubin-total are in units per liter.
  there were no difference in each group.
Kidney function | at the start of the experiment and at the 4th, 10th week
  Serum BUN,Creatine and urine acid are in milligram per deciliter
  there were no difference in each group.
Lipid profile | at the start of the experiment and at the 4th, 10th week
  Serum HDL-Cho, LDL-Cho, triglyceride and total cholesterol are in milligram per deciliter
  there were no difference in each group.
Hematology | at the start of the experiment and at the 4th, 10th week
  Serum WBC in 1000/uL , RBC in 1000000/uL, hemoglobin in gram per deciliter, hematocrit in percentage , MCV in femtoliter , MCH in picogram, MCHC in gram per deciliter, platelet in 1000/uL ; neutrophils, lymphocytes, monocytes, eosinophils and basophils are in percentage.
  there were no difference in each group.
Iron status | at the start of the experiment and at the 4th, 10th week
  Serum iron, ferritin and TIBC are in microgram per deciliter
  there were no difference in each group.
Antioxidative status | at the start of the experiment and at the 4th, 10th week
  Thiobarbituric acid-reactive substance, glutathione/oxidized glutathione ratio ,and plasma 8-isoprostane.
  During PE supplementation, plasma TBARS level was significantly lower than placebo group (p < 0.05), and there was no significant difference between baseline and PE group.
  During PE supplementation, GSH / GSSG ratio in red blood cells was significantly higher than baseline and placebo group (p < 0.05), but there was no significantly difference between baseline and placebo group.
  After 4 weeks of supplementation PE and Placebo, the results of plasma 8-isoprostane level were shown in Figure 7C. There was no significantly difference in each group.
Food frequency questionnaire | at the beginning, 4th, 7th and 10th of the experiment
  To analyze nutrition status of participants.
  the frequency of staple foods, vegetables, fruits and milk intake insufficient in one day.
Three-day dietary record. | at 2nd , 4th, 6th and 10th week of study
  To analyze nutrition status of participants.
  The intake of carbohydrates and fat of three major nutrients was insufficient and protein was excessive.
  In terms of vitamins, vitamin B1, vitamin B2, vitamin E consumed appropriately, vitamin B6, vitamin A consumed excessively, Vitamin C was insufficient.
  In micronutrients, calcium and iron was insufficient, and sodium, zinc and magnesium consumed in moderation.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Taiwan Adventist Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No